CLINICAL TRIAL: NCT05821842
Title: Sonu Nasal COngestion RElief Study (SCORE)
Brief Title: Sonu Nasal Congestion Relief Study in Patients Suffering From Moderate to Severe Nasal Congestion
Acronym: SCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Wave Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP-002
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-09

CONDITIONS: Nasal Congestion and Inflammations
MeSH Terms: conditions — Nasal Obstruction; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Sonu Treatment Group (Experimental): Patients will receive acoustic resonance therapy for 15 minutes, twice a day, for two weeks using Sonu.
  Interventions: Device: Sonu
- Sham Control Group (Sham Comparator): Patients will receive non-resonant acoustic energy for 15 minutes, twice a day, for two weeks using Sonu.
  Interventions: Device: Sonu

INTERVENTIONS:
Device: Sonu — Acoustic energy delivery

SUMMARY:
To demonstrate the safety and effectiveness of Sonu for the treatment of patients suffering from moderate to severe nasal congestion.

DETAILED DESCRIPTION:
Sonu consists of and acoustic vibrational headband worn circumferentially at the level of the forehead. A smart phone App, paired to the headband, delivers acoustic resonant frequencies of the subject's nasal cavity through the headband and provides relief. Sonu is intended to be used for the treatment of moderate to severe nasal congestion due to rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Present with symptoms of nasal congestion for 1 month or more prior to treatment
* Have a 24 hour reflective nasal congestion subscore of the TNSS of 2 or more on a 0 to 3 scale at the time of screening

Exclusion Criteria:

* Head, nasal or sinus surgery within 3 months
* Sinus infection diagnosed within the last month, or rhinitis medicamentosa
* Documented history of nasal polyposis or mass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Johnson, MD, Principal Investigator — San Francisco Otolaryngology Medical Group
Locations (1):
- San Francisco Otolaryngology Medical Group, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 66 subjects were screened and 52 subjects were enrolled between March 2022 and May 2023 at 3 sites.
Groups:
- Sonu Treatment Group: Patients will receive acoustic resonance therapy for 15 minutes, twice a day, for two weeks using Sonu.
  Sonu: Resonance acoustic energy delivery
- Sham Control Group: Patients will receive non-resonant acoustic energy for 15 minutes, twice a day, for two weeks using Sonu.
  Sonu: Non-resonance acoustic energy delivery
Period: Overall Study
Arm/Group | Sonu Treatment Group | Sham Control Group
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sonu Treatment Group | Sham Control Group | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (17.7) | 48.8 (14.9) | 47.1 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 30
  Male | 16 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 20 | 22 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 17 | 31
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 5 | 5 | 10
Nasal Congestion Sub-score [Mean (Standard Deviation); unit: units on a scale of 0-3] — Nasal congestion sub-score is reported on using a scale of 0-3 based on the severity of nasal congestion symptoms (0=None, 1=Mild, 2=Moderate, or 3=Severe). 0 is the minimum and 3 is the maximum. Higher scores mean worse outcomes.
  units on a scale of 0-3 | 2.27 (0.45) | 2.12 (0.33) | 2.20 (0.39)

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness
Description: Change in nasal congestion sub-score compared to baseline. The nasal congestion sub-score is reported on a scale of 0-3. 0 is the minimum and 3 is the maximum. Higher scores mean worse outcomes.
Time Frame: 2 weeks
Population: Adults (18 years of age or and older) suffering from moderate to severe nasal congestion from rhinitis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sonu Treatment Group | Sham Control Group
Number analyzed (Participants) | 26 | 26
score on a scale | -0.87 [-1.11 to -0.62] | -0.44 [-0.64 to -0.23]

2. Secondary Outcome: Secondary Effectiveness
Description: Change in total nasal symptom score (TNSS) compared to baseline. The TNSS is the sum of four (4) symptom sub-scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, each self-rated by the subject using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe. TNSS scores are reported on a scale of 0-12. 0 is the minimum and 12 is the maximum. Higher scores mean worse outcomes.
Time Frame: 2 weeks
Population: Adults (18 years of age or older) suffering from moderate to severe nasal congestion from rhinitis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sonu Treatment Group | Sham Control Group
Number analyzed (Participants) | 26 | 26
score on a scale | -2.85 [-3.85 to -1.85] | -1.32 [-2.27 to -0.36]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Sonu Treatment Group | Sham Control Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT05821842/Prot_SAP_000.pdf